CLINICAL TRIAL: NCT07157059
Title: Labor and Delivery Doula Program to Reduce Perinatal Morbidity and Mortality in Kansas
Acronym: Doula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: BioNexus KC (Unknown); Blue KC (Blue Cross Blue Shield) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00161314; FP00000002 (Other Grant/Funding Number: BioNexus KC); IRB STUDY00149318 (Other: The University of Kansas Medical Center)
Record Dates: First submitted 2025-08-18; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related; Doula Care; Black Maternal and Infant Health; Prenatal Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doula-Enhanced Care Group (Experimental): This group received doula-enhanced care along with routine pregnancy care.
  Interventions: Behavioral: Doula Care
- Routine Pregnancy Care Group (No Intervention): This group received routine pregnancy care.

INTERVENTIONS:
Behavioral: Doula Care — Participants assigned to the Doula care group received care from the doula pre, during, and post delivery.
  Arms: Doula-Enhanced Care Group

SUMMARY:
The study was done to learn how doula-enhanced care provided to Black birthing people improved perceived communication and quality care.

ELIGIBILITY:
Inclusion Criteria:

* Black birthing people
* Received care and plan to delivery at the University of Kansas Medical Center
* Scored positive to social determinants of health screener
* Gestational age between 14-27.6 weeks at enrollment

Exclusion Criteria:

* Pregnancy not viable or pregnancy not intrauterine on ultrasound
* Patients who are not willing to be randomized into not receiving doula enhanced
* Patients who do not plan to delivery at the University of Kansas Health System
* Non-Black birthing people.
* Planned cesarean section
* Patients with a known major fetal anomaly
* Non-English speaking

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Perceptions of provider communication | 14-28 weeks GA through 6-weeks postpartum
  Assess perceptions of provider communication using Likert-scale surveys (including some yes/no questions and comments).
Perceptions of maternal care | 14-28 weeks GA through 6-weeks postpartum
  Assess perceptions of maternal care using Likert-scale surveys (including some yes/no questions and comments).

SECONDARY OUTCOMES:
Perinatal outcome - gestational age (GA) at delivery | 14-28 weeks GA through delivery
  Assess gestational age (GA) at delivery by collecting data from their patient surveys and chart.
Perinatal outcome - preterm <37 weeks births | 14-28 weeks GA through delivery
  Assess preterm <37 weeks births by collecting data from their patient surveys and chart.
Perinatal outcome - cesarean sections | 14-28 weeks GA through delivery
  Assess cesarean sections by collecting data from their patient surveys and chart.
Perinatal outcome - gestational hypertension/Preeclampsia | 14-28 weeks GA through delivery
  Assess gestational hypertension/Preeclampsia by collecting data from their patient surveys and chart.
Neonatal morbidity | Birth through 6-weeks postpartum
  Assess neonatal morbidity by collecting neonatal APAGAR scores and neonatal ICU admissions
Antepartum depression | 14-28 weeks GA through delivery
  Assess depression using Edinburgh depression screening tool
Postpartum depression | Birth (delivery) through 6-weeks postpartum
  Assess depression using Edinburgh depression screening tool
Maternal pain management | Birth through 6-weeks postpartum
  Assess pain management via postpartum pain perception scores and total morphine milliequivalent used.
Lactation Status | Birth through 6-weeks postpartum
  Assess lactation status was asked and recorded for patients during their labor and delivery admission and postpartum visits

CONTACTS AND LOCATIONS:
Overall Officials: Angela Martin, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States